CLINICAL TRIAL: NCT04912674
Title: Prospective Evaluation of Symphony™ Posterior Cervical System for Surgical Treatment of Adult Cervical Deformity: A Multi-Center Study
Brief Title: Evaluation of Symphony™ Posterior Cervical System for Surgical Treatment of Adult Cervical Deformity
Acronym: Symphony
Status: Recruiting | Type: Observational
Sponsor: International Spine Study Group Foundation (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Other Study IDs: 2140
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cervical Deformity
Keywords: Cervical deformity; Kyphosis; Scoliosis
MeSH Terms: conditions — Kyphosis; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Operative: Inclusion Criteria:
  1. ≥18 years old at time of treatment
  2. Patient undergoing a posterior cervical instrumented fusion using the DePuy Synthes SymphonyTM OCT System for the treatment of adult cervical deformity, defined as any of below criteria:
     1. Loss of cervical lordosis (≤ 0° cervical lordosis C2-7)
     2. ≥ 5° of kyphosis across any 1 or 2 cervical segments
     3. ≥ 10° of cervical scoliosis
     4. C2-C7 SVA ≥ 4cm
     5. T1 Slope minus Cervical Lordosis ≥ 20°
     6. Grade I or greater Spondylolisthesis at any segment C1-T1
     7. Horizontal Gaze ≤ 0 or ≥ 11
  3. Plan for surgical correction of cervical deformity in the next 6 months
  4. Willing to provide consent and complete study forms at baseline and follow-up intervals
  Exclusion Criteria:
  1. Active spine tumor or infection
  2. Deformity due to acute trauma
  3. Unwilling to provide consent or to complete study forms
  4. Prisoner
  5. Pregnant or immediate plans to get pregnant
  Interventions: Device: Symphony OCT System

INTERVENTIONS:
Device: Symphony OCT System — Surgical intervention will be patient specified by treating surgeon.

SUMMARY:
Multi-center, prospective, non-randomized study to evaluate Symphony™ Posterior Cervical System in the setting of surgical treatment of adult cervical deformity.

DETAILED DESCRIPTION:
Specific Aims:

* Evaluate outcomes for operative treatment of adult cervical deformity patients treated with posterior spinal fusion using SymphonyTM posterior cervical system at 6 weeks, 1 year, and 2 year follow up. Outcome metrics will include standardized patient reported outcome measures, radiographic analysis of deformity correction and spinal alignment.
* Evaluate rates and risk factors for perioperative complications and need for revision surgery at 6 weeks, 1 year, and 2 years postoperatively.
* Develop and validate a surgical invasiveness index for cervical deformity surgical procedures
* Validate the cervical deformity frailty index previously developed by the ISSG and further optimize this index
* Establish adult cervical deformity specific thresholds for minimal clinically important difference (MCID) for standard outcomes measures using a patient satisfaction anchor
* Develop a series of predictive models for adult cervical deformity surgery, including outcomes (e.g. overall change and achievement of MCID), occurrence of complications, and radiographic changes
* Assess the psychological impact of adult cervical deformity, how psychological measures change following surgical treatment, and whether there are correlations between baseline psychological factors and outcomes following surgery
* Assess baseline functional measures (e.g. grip strength) for adult cervical deformity patients presenting for surgery, assess how these functional measures change following surgery, and assess whether there are correlations between baseline functional measures and likelihood to improve following surgery
* Assess baseline narcotic use among adult cervical deformity patients presenting for surgery
* Assess changes in narcotic use from baseline to follow-up intervals after surgical treatment for adult cervical deformity
* Assess for correlations between narcotic use (baseline and follow-up) and outcomes following surgical treatment for adult cervical deformity
* Assess the impact of osteopenia and osteoporosis on patient frailty, complications, and maintenance of deformity correction
* Define clinical and demographic features of the population afflicted with cervical deformity (e.g., age, gender, comorbidities, disability, health-related quality of life)
* Assess for correlations between radiographic parameters and degree of disability/pain at baseline
* Assess and describe surgical strategies used to address cervical deformity
* Define complications and rates of complications (perioperative and delayed) associated with the surgical treatment of cervical deformity
* Assess the role/need for pre/post operative tracheostomy and PEG
* Evaluate and compare radiographic changes of sagittal spinal alignment (focal, regional, and global) and pelvic parameters pre and post cervical deformity surgery.
* Develop predictive formulas of post-operative alignments based on surgical techniques employed for correction
* Identify risk factors related to poor clinical outcomes
* Define potential impact of complications on clinical/radiographic outcomes
* Determine reoperation rates over two-year follow-up period
* Assess change in subaxial alignment after occiput to C2 fusion
* Assess the effect of C1-2 lordosis and C1-2 fusion on subaxial alignment and outcome
* Assess outcomes of long fusions involving the occiput related to head center of gravity and regional and global balance
* Assess outcomes of occipital-cervical-thoracic fusion on cervical alignment and global alignment
* Evaluate clinical outcomes (short- and long-term) following cervical deformity surgery
* Assess cost-effectiveness of adult cervical deformity surgery
* Correlate different measures of frailty, including Edmonton, CHSA, and ISSG.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old at time of treatment
2. Patient undergoing a posterior cervical instrumented fusion using the DePuy Synthes SymphonyTM OCT System for the treatment of adult cervical deformity, defined as any of below criteria:

   1. 10 degrees of overall cervical kyphosis (measured from C2-C7)
   2. 10 degrees of kyphosis across any 1 or 2 cervical segments
   3. 10 degrees of scoliosis
   4. C2-C7 SVA >4cm
3. Plan for surgical correction of cervical deformity in the next 6 months
4. Willing to provide consent and complete study forms at baseline and follow-up intervals

Exclusion Criteria:

1. Active spine tumor or infection
2. Deformity due to acute trauma
3. Unwilling to provide consent or to complete study forms
4. Prisoner
5. Pregnant or immediate plans to get pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cervical deformity patients from spine surgeon clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2027-07-12 (Estimated); Study Completion 2027-07-12 (Estimated)

PRIMARY OUTCOMES:
Pain Numeric rating scale (NRS) - Headaches | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Self reported pain in Head where 0=no pain/10=severe pain
Pain Numeric rating scale (NRS) - Neck | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Self-reported pain in Neck where 0=no pain/10=severe pain
Pain Numeric rating scale (NRS) - Upper extremity | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Self-reported pain in Arms where 0=no pain/10=severe pain
Pain Numeric rating scale (NRS) - Lower extremity | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Self-reported pain in Legs where 0=no pain/10=severe pain
Pain Numeric rating scale (NRS) - Back | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Self-reported pain in Back where 0=no pain/10=severe pain
Neck Disability Index (NDI) | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Patient reported neck disability tool
Veterans RAND 12 Item Health Survey (VR-12) | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Anxiety | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Depression | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Pain Interference | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Physical Function | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Satisfaction (Role) | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Computer adaptive PROs
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Satisfaction (DSA) | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Computer adaptive PROs
Spine Radiographs | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Radiographic parameters (Cervical lordosis, Kyphosis, Scoliosis; Global balance in coronal and sagittal planes of the spine; pelvic parameters (pelvic incidence, tilt, slope) and bony fusion status
Modified Japanese Orthopaedic Association Scale (mJOA) | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Patient reported outcome measuring functional status using scale of 0 to 18. The higher the score, the less disability.

SECONDARY OUTCOMES:
EAT-10 | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Measures swallowing difficulties as reported by the patient.
Voice Handicap Index (VHI-10) | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Measures voice handicap as reported by the patient.
Adverse events | 6 weeks, 1 year, and 2 years
  Any adverse events that occur during study participation & meeting study established reporting criteria
Edmonton Frail Scale | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Frailty scale from 0 to 17 where the higher the score the more frail the patient
CHSA Frail Scale | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  Clinical Frailty Scale from 1 to 9 where the higher the score, the more frail the patient
Dynamometer Hand Grip Strength test | Change from Preop to 6 weeks, 6 months, and 1 & 2 year follow-up
  With patient seated, patient will squeeze the dynamometer as hard as he/she can with each hand.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Smith, MD, PhD, Principal Investigator — University of Virginia; Christopher Shaffrey, MD, Principal Investigator — Duke University; Shay Bess, MD, Principal Investigator — Denver Int'l Spine Center, Rocky Mountain Hospital for Children & Presbyterian St. Luke's MC
Locations (7):
- United States (7):
  - University of California Davis, Sacramento, California
  - Denver International Spine Center, Rocky Mountain Hospital for Children and Presbyterian St. Luke's Medical Center, Denver, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No